CLINICAL TRIAL: NCT06607991
Title: Study of Blinatumomab for the Treatment of Calcineurin Inhibitor-Resistant or Intolerant Steriod-Resistant Nephrotic Syndrome in Pediatric Patients
Brief Title: Blinatumomab for CNI-Resistant/Intolerant SRNS in Children
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IRB-0241-P-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: CNI-resistant Steriod Resistant Nephrotic Syndrome; CNI-intolerent; Steriod Resistant Nephrotic Syndrome; Multidrug Resistant Nephrotic Syndrome
Keywords: CNI-resistant SRNS; children; Blinatumomab; Multidrug resistant steroid resistant nephrotic syndrome; steroid resistant nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab Treatment (Experimental)
  Interventions: Drug: Blinatumomab Treatment

INTERVENTIONS:
Drug: Blinatumomab Treatment — Blinatumomab treatment for CNI-resistant/Intolerant pediatric steriod-resistant nephrotic syndrome Patients will receive two 5-day cycles of Blinatumomab (5 µg/m²/day, maximum dose 9 µg/day), administered intravenously. The second cycle will begin on the first day of the third week following the first cycle.

SUMMARY:
This exploratory clinical trial aims to evaluate the efficacy and safety of Blinatumomab in treating children with calcineurin inhibitor (CNI)-resistant or multidrug-resistant steroid-resistant nephrotic syndrome (SRNS). Eligible participants include pediatric patients aged 2 to 17 years who have either failed to respond to adequate CNI therapy or are resistant to at least two classes of immunosuppressants, including CNIs and biologics. A short course of low-dose Blinatumomab will be administered in an open-label, single-arm, self-controlled trial design. The study seeks to determine whether Blinatumomab can reduce proteinuria and induce clinical remission in this difficult-to-treat population, offering a potential new therapeutic option for children with limited response to conventional therapies.

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) in children is characterized by excessive proteinuria, hypoalbuminemia, hyperlipidemia, and edema. Approximately 15-20% of pediatric NS cases are classified as steroid-resistant nephrotic syndrome (SRNS), a condition associated with poor prognosis and limited response to standard therapies. Calcineurin inhibitors (CNIs) are frequently used as first-line immunosuppressants in SRNS; however, a subset of patients demonstrate resistance to or intolerance of CNIs. Moreover, a proportion of patients may be refractory to multiple classes of immunosuppressive agents, including biologics, posing a significant therapeutic challenge.

This exploratory, single-center, open-label clinical trial is designed to evaluate the safety and efficacy of Blinatumomab-a bispecific T-cell engager targeting CD19-positive B cells-in pediatric patients with CNI-resistant or multidrug-resistant SRNS. Eligible participants will include children aged 2 to 17 years who have either not responded to adequate CNI therapy or have failed to achieve remission despite treatment with at least two classes of immunosuppressive agents (including CNIs and biologics).

A total of 6 patients will be enrolled and administered two short courses of low-dose Blinatumomab intravenously, each lasting 5 days. The primary efficacy outcome will be the rate of complete or partial remission of proteinuria. Secondary outcomes will include safety and tolerability assessments, changes in immunologic markers, and renal function monitoring. By selectively depleting CD19-positive B cells, Blinatumomab may modulate aberrant immune activation that underlies treatment-resistant SRNS.

This study seeks to generate preliminary data on the potential therapeutic role of Blinatumomab in this difficult-to-treat pediatric population, with the ultimate goal of identifying a novel immunomodulatory approach for SRNS patients with limited treatment options.

ELIGIBILITY:
- Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1.Age between 2 and 17 years, regardless of gender. 2.Meet the 2021 KDIGO definition of steroid-resistant nephrotic syndrome (SRNS), and fulfill either of the following:

1. Have received an adequate dose of calcineurin inhibitors (CNIs) for more than 6 months without achieving at least partial remission.
2. Or have contraindications to CNI use, including:

1) Significant renal impairment, defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m², or presence of acute kidney injury at the time of diagnosis; 2) Renal biopsy showing prominent acute or chronic tubular injury, such as tubular atrophy or interstitial fibrosis involving more than 50% of the sampled tissue; 3) Elevated urinary markers (β2-microglobulin, α1-microglobulin, or retinol-binding protein) exceeding three times the upper limit of normal; 4) Abnormal glucose tolerance; 5) Severe uncontrolled hypertension, defined as systolic and/or diastolic blood pressure ≥ the 95th percentile + 12 mmHg for age, sex, and height, or ≥ 140/90 mmHg; 6) Concomitant use of medications known to have significant interactions with CNIs, leading to increased toxicity or reduced efficacy; 7) Known allergy or hypersensitivity to CNIs or any of their components. (3) Or have demonstrated inadequate response or disease relapse after treatment with at least two immunosuppressive agents, including CNIs and at least one of the following:

1. Conventional immunosuppressive agents: cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide
2. Biologic agents: abatacept, ofatumumab, obinutuzumab, rituximab Inadequate response is defined as failure to achieve complete remission after 12 months of therapy or relapse following initial response.

3. Renal biopsy performed prior to screening confirms a diagnosis of minimal change disease (MCD) or focal segmental glomerulosclerosis (FSGS).

4. The subject and/or their legal guardian must provide written informed consent, indicating understanding of the study's purpose and procedures, with the right to withdraw consent at any time without affecting the subject's future medical care.

-Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. eGFR < 60 mL/min/1.73 m² (using the modified Bedside Schwartz formula);
2. Stroke or seizure within 6 months prior to screening, or other active central nervous system disorders;
3. Genetic nephropathy confirmed by genetic testing;
4. Renal biopsy confirming IgA nephropathy, membranous nephropathy, or membranoproliferative glomerulonephritis;
5. Severe congenital heart disease or history of acute myocardial infarction within 6 months, or severe arrhythmias (e.g., frequent multifocal ventricular or supraventricular tachycardia, ventricular tachycardia), or moderate to large pericardial effusion, severe myocarditis, or unstable vital signs requiring vasopressors to maintain blood pressure;
6. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with hepatitis B virus (HBV) DNA levels above the normal range; positive for hepatitis C virus (HCV) antibodies with HCV RNA levels above the normal range; or positive for human immunodeficiency virus (HIV) antibodies, syphilis, or cytomegalovirus (CMV) DNA;
7. Abnormal laboratory values prior to screening: moderate to severe neutropenia (≤1.0×10⁹/L); moderate to severe anemia (hemoglobin ≤90 g/L); thrombocytopenia (≤75×10⁹/L); or liver dysfunction (ALT, AST, or bilirubin greater than 2.5 times the upper limit of normal and persisting for 2 weeks);
8. Subjects with tumors or other life-threatening diseases prior to screening;
9. Positive blood pregnancy test;
10. Participation in other clinical trials within 1 month prior to enrollment;
11. Received rituximab or cyclophosphamide therapy within the past 3 months;
12. Any other condition deemed by the investigator to be unsuitable for participation;
13. Vaccination with live vaccines within 4 weeks prior to screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-09-19 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and safety of Blinatumomab | with 24 weeks of Blinatumomab treatment
  Effectiveness: The primary endpoint is the proportion of patients achieving complete or partial remission within 24 weeks of treatment. Complete remission is defined as a urinary protein/creatinine ratio (UPCR) ≤ 200 mg/g for three consecutive days, while partial remission is defined as a ≥ 50% reduction in proteinuria from baseline with a UPCR between 200 and 2000 mg/g.
  Safety: Adverse events (AEs) and serious adverse events (SAEs) will be monitored and classified according to the CTCAE v5.0. This includes events such as cytokine release syndrome, fever, headache, and potential neurotoxicity.

SECONDARY OUTCOMES:
long-term efficacy of Blinatumomab and Immunological Markers | with 52 weeks of Blinatumomab
  Secondary Outcome Measures:
  Long-term Efficacy: Maintenance of remission at 52 weeks will be evaluated, along with the time to remission and the duration of remission.
  Immunological Markers: Changes in CD19+ B cell counts, particularly depletion and subsequent recovery of B cell populations, will be monitored.
  Recurrence of Disease: The time to first relapse and the proportion of patients who relapse during the 52week follow-up period will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, PhD, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No